CLINICAL TRIAL: NCT05083416
Title: Effect of Prolonged Nightly Fasting (PNF) on Immunotherapy Treatment Outcomes in Patients With Advanced Head and Neck Cancer (HNSCC)-Role of Gut Microbiome
Brief Title: Effect of Prolonged Nightly Fasting on Immunotherapy Outcomes in HNSCC - Role of Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-21150; 20121102 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2021-10-04; First posted 2021-10-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer
Keywords: Intermittent Fasting
MeSH Terms: conditions — Head and Neck Neoplasms; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Prolonged Nightly Fasting (Experimental): Participants will be educated on Prolonged Nightly Fasting (PNF) and the "mycircadianapp". Participants be allowed to choose any 10-hr period that falls between 6 AM- 6 PM, as feeding period. Participants will be recommended to follow study diet guidelines, eat to satiety and not count calories. Participants will be allowed to have water, beverages (<4 kcal) during the fasting period.
  Interventions: Behavioral: Prolonged Nightly Fasting
- B: Regular Eating pattern (Active Comparator): Participants will follow a traditional eating pattern with no time restrictions.
  Interventions: Behavioral: Regular Eating pattern

INTERVENTIONS:
Behavioral: Prolonged Nightly Fasting — Limiting daily period of food intake to 10 hours and nightly fasting period to 14 hours.
  Other Names: Intermittent Fasting
  Arms: A: Prolonged Nightly Fasting
Behavioral: Regular Eating pattern — Food intake not limited to a specific time during day/night.
  Arms: B: Regular Eating pattern

SUMMARY:
This study aims to evaluate if eating within an 8-10-hour window during the day, without any caloric restriction, can lead to better response rates to immunotherapy in head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed recurrent /metastatic head and neck squamous cell cancer that is not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy) and initiating standard of care immune checkpoint blocker- (Nivolumab, pembrolizumab, Atezolizumab, Avelumab or Durvalumab with or without chemotherapy), for the first time.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

Exclusion Criteria:

* BMI< 18.5.
* Diabetes mellitus, hyperthyroidism, pregnancy, any eating disorder including anorexia nervosa or bulimia, metabolic disorders that may affect gluconeogenesis or adaptation to short fasting periods
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disease requiring systemic steroids, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have known leptomeningeal metastases or untreated or symptomatic brain metastases. Treated, asymptomatic brain metastasis can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Rates of Prolonged Nightly Fasting (PNF) compliance | at 3 months
  Adherence to the 8-10 hour time restricted feeding window will be measured using "mycircadianclock" app ,which has been validated as a tool to conveniently and reliably track time of food intake and its correlation with timing of the day and sleep. It can be tailored to restrict feeding duration to specific set points.
Change in gut microbiome and microbial metabolites | Baseline and at 12 weeks
  Changes in gut microbiome composition/diversity as well as gut microbial metabolites in participants using PNF will be compared with participants that are not restricting eating times will be measured using stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No